CLINICAL TRIAL: NCT00473824
Title: A Randomized, Open-Label Phase II Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Hepatitis C Immune Globulin Intravenous (Human), Civacir(TM), in Liver Transplant Recipients
Brief Title: Randomized Phase II Study of Hepatitis C Immune Globulin Intravenous (Human), Civacir(TM), in Liver Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: New sponsor's decision to pursue a redesigned clinical study
Sponsor: ADMA Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nabi-3104
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Sequelae of Viral Hepatitis; Transplantation Infection; Evidence of Liver Transplantation
Keywords: hepatitis C; liver transplantation; immune globulin
MeSH Terms: conditions — Hepatitis C | interventions — hepatitis C immune globulin, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Civacir Treated (Experimental): Hepatitis C Immune Globulin Intravenous (Human) 5% [Civacir], 18 infusions total, per schedule, of Civacir 300 or 400 mg/kg of body weight, with standard post-transplant site specific routine immunosuppressant therapy .
  Interventions: Biological: Hepatitis C Immune Globulin Intravenous (Human) 5%
- Observational Control (No Intervention): Observation on standard post-transplant site specific routine immunosuppressant therapy without infusions of Hepatitis C Immune Globulin Intravenous (Human) 5% [Civacir].

INTERVENTIONS:
Biological: Hepatitis C Immune Globulin Intravenous (Human) 5% — Hepatitis C Immune Globulin Intravenous (Human) 5%, [Civacir]: 18 infusions total, per schedule, of 300 or 400 mg/kg of body weight given with standard post-transplant therapy inclusive of immunosuppressive agents.
  Other Names: Civacir™
  Arms: Civacir Treated

SUMMARY:
A Phase 2 study to evaluate safety, pharmacokinetics and efficacy of Hepatitis C Immune Globulin Intravenous (human) [Civacir(TM)] for preventing or reducing the impact of recurrent HCV infection following liver transplantation.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is the leading single cause of liver transplantation (LT) in the US and Europe. Recurrence of HCV infection following LT is almost universal. There is currently no effective way to prevent post-transplantation HCV infection of the liver graft and related progression of HCV-related liver disease. This study is designed to evaluate a polyclonal human hepatitis C immune globulin (Civacir) given during and post liver transplantation for preventing or reducing the impact of recurrent HCV infection.

In this open-label trial, 2 subjects will be randomized to receive Civacir (standard of care treatment plus Civacir) for every 1 Control subject (standard of care treatment alone). Civacir recipients will receive 18 intravenous infusions over 24 weeks beginning at the time of liver transplantation.

Viral loads, liver enzyme assessments and liver biopsy assessments will be made at scheduled intervals during the study which will last for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age.
* Written informed consent.
* Expectation of compliance with the protocol procedures.
* If female, have a negative pregnancy test within 3 days prior to randomization and use an acceptable method of contraception or be at least one year post-menopausal or surgically sterile.
* HCV infection identified by positive, quantifiable HCV-RNA test within 3 months prior to transplantation.
* First time liver transplant recipient.
* Primary, single organ recipient (deceased donor <65 years of age).
* Normal TSH.
* Subjects with a pre-LT diagnosis of hepatocellular carcinoma (HCC) may be enrolled provided: there is no evidence of extrahepatic spread, tumor is solitary and <5cm or there are up to three tumors <3 cm.
* Agree to receive study medication as outlined in the protocol and follow all study related procedures until the conclusion of their protocol participation.
* Agree to consume no alcohol during the entire study period.

Exclusion Criteria:

* Has received an investigational agent within the last six weeks prior to liver transplantation. Exceptions include Theraspheres for hepatocellular carcinoma or rifaximin.
* Known immunoglobulin A deficiency.
* Subject weighs more than 112.5 Kg (248 pounds).
* Known history of cancer, suspected cancer, or cancer therapy within 12 months prior to the administration of the investigational product, except for treatment for basal cell carcinoma, squamous cell carcinoma, cancer of the cervix in situ, early stage prostate cancer (Gleason's grade 1 or 2), or a history of malignancy where the risk of recurrence is >= 20% within 2 years. A significant exception is hepatocellular carcinoma with predefined acceptability (see inclusion criteria).
* Has any condition judged by the study physician to preclude participation in the study, including any psychological disorder, which might hinder compliance.
* History of use of immunosuppressive or immunomodulatory drugs within 3 months prior to randomization (except low-dose physiologic replacement glucocorticoid therapy (<=10 mg of prednisone or equivalent per day).
* Recipient of liver from a living donor.
* Subjects whose liver is obtained from a non-beating heart donor.
* Subjects scheduled to receive a split liver transplantation.
* Liver transplants that were obtained from donors across ABO incompatible blood type.
* Donor liver cold ischemic time greater than 20 hours.
* Donor liver is from a hepatitis C positive donor.
* Evidence of any other unresolved infection and any unresolved opportunistic infection requiring treatment.
* Serum creatinine level >2.0 times the upper limit of normal or advanced renal disease at screening.
* Neutrophil count <1500 cells/mm3, WBC>20,000 x 109/L, Hgb <8 g/dL, or platelet count <25,000 cells/mm3.
* Planned use of T-cell depleting antibody therapies.
* Hepatitis B (sAg, cAb IgM), hepatitis A (IgM) or HIV infection.
* History of autoimmune disease (SLE, scleroderma, RA, etc.).
* Women who are pregnant or breast feeding.
* The use of colony stimulating factor agents to facilitate subject's entry into study within 2 weeks of enrollment.
* History of severe psychiatric disease, especially depression.
* Seizure disorders uncontrolled by anticonvulsants (within the last 12 mos).
* History of severe cardiac disease, unhealed gastric or duodenal ulcer, or other significant medical disease that would put the subject at risk from the volume of the infusions or significant risk of bleeding from the underlying condition.
* Evidence of alcohol and/or drug abuse within 6 months of entry or inability/unwilling-ness to abstain from alcohol throughout entire course of treatment and follow-up.
* Concomitant medication with rifabutin, pyrazinamide, isoniazid, thalidomide, oxymetholone (Anadrol).
* History of thyroid disease poorly controlled on prescribed medications.
* History or other evidence of severe illness or any other conditions which would make the subject, in the opinion of the investigator, unsuitable for Civacir treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Katz, MD, Study Director — Clinical Trial and Consulting Services; Shailesh Chavan, MD, Study Director — Biotest Pharmaceuticals
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First enrollment: 14 May 2007 Last Subject completed: 16 February 2009 Three investigative sites, all Mayo Clinics
Pre-assignment Details: This was an open label, randomized study.
Groups:
- Civacir Treatment Arm: Subjects received standard site specific routine post-transplant immunosuppressant therapy with Hepatitis C Immune Globulin Intravenous (Human) 5% [Civacir], 18 infusions total, per schedule, of Civacir 300 or 400 mg/kg of body weight.
- No Civacir (Control): Observation on standard site specific routine post-transplant immunosuppressant therapy without infusions of Hepatitis C Immune Globulin Intravenous (Human) 5%.
Period: Overall Study
Arm/Group | Civacir Treatment Arm | No Civacir (Control)
Started | 5 | 2
Completed | 0 (Study Completion/Early Termination Date) | 2 (Study Completion/Early Termination Date)
Not Completed | 5 | 0
Not completed — Virologic Breakthrough | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by physician | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Civacir Treatment Arm | No Civacir (Control) | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (5.0) | 47 (11.3) | 50 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Post Transplant Reduction in Viral Load (as Measured Quantitatively by Hepatitis C Virus (HCV) Reverse Transcription-Polymerase Chain Reaction (HCV RT-PCR)).
Description: Percentage of subjects who achieve reduction in viral load from the baseline pre-transplant value. Baseline is the pre-transplant HCV viral load as measeured by RT-PCR. Post-transplant HCV viral load is determined at both 1 month and 6 months post-tranplant.
Time Frame: Outcome evaluations at 1 month (Day 28) and 6 months ( 24 weeks) post-tranplant.
Population: As the study was terminated early and since no participant in either arm achieved reduction in viral load, it was recorded that zero particpants and zero percent in each arm achieved reduction in viral load.
Measure: Number; unit: percentage of participants
Groups:
- Civacir Treatment Arm: Subjects received Hepatitis C Immune Globulin Intravenous (Human) 5% [Civacir], 18 infusions total, per schedule, of Civacir 300 or 400 mg/kg of body weight, in addition to their standard site specific routine post-tranplant immunosuppressant therapy.
- No Civacir (Control): Observation on standard site specific routine post-tranplant immunosuppressant therapy without infusions of Hepatitis C Immune Globulin Intravenous (Human) 5%. Standard post-tranplant therapy includes immunosuppressive agents.
Arm/Group | Civacir Treatment Arm | No Civacir (Control)
Number analyzed (Participants) | 5 | 2
percentage of participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Civacir Treatment Arm | No Civacir (Control)
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/2
Other Adverse Events (participants affected / at risk) | 4/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Civacir Treatment Arm (N=5) | No Civacir (Control) (N=2)
Adult Respiratory Distress Syndrome [ARDS] (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest Tightness (General disorders) | 1 (1) | 0 (0)
Mid Common Hepatic Ductal Stricture with possible Biliary Leak (Surgical and medical procedures) | 1 (1) | 0 (0)
Vancomycin-Resistant Enterococcus Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Methicillin-resistant staph aureus (MRSA) Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalemia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Civacir Treatment Arm (N=5) | No Civacir (Control) (N=2)
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 1 (1) | 0 (0)
Eye Disorders (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 3 (14) | 2 (8)
General Disorders and Administration Site Conditions (General disorders) | 3 (3) | 1 (4)
Hepatobiliary Disorders (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infections and Infestations (Renal and urinary disorders) | 1 (2) | 1 (1)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Investigations (Investigations) | 0 (0) | 1 (1)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 3 (6) | 2 (4)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
Nervous System Disorders (Nervous system disorders) | 2 (4) | 2 (3)
Psychiatric Disorders (Psychiatric disorders) | 3 (3) | 2 (4)
Renal and Urinary Disorders (Renal and urinary disorders) | 1 (2) | 2 (2)
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vascular Disorders (Vascular disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination by sponsor due to data from the initial 7 patients of 36 planned for this study. Therefore, statistical analysis was not performed and no conclusion were reached regarding efficacy or drug safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less